CLINICAL TRIAL: NCT01733030
Title: The Effects of D-cycloserine on Stimulus Generalization of Conditioned Fear in Healthy Controls.
Brief Title: The Effects of D-cycloserine on Stimulus Generalization of Conditioned Fear Healthy Controls.
Acronym: DCS
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: MH080130
Record Dates: First submitted 2012-11-19; First posted 2012-11-26 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Post Traumatic Stress Syndrome
Keywords: PTSD
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic | interventions — Cycloserine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 250 mg Seromycin: Healthy adults who will receeve one administration of 250 mg of Seromycin prior to the start of the study.
  Interventions: Drug: Seromycin
- 500 mg Seromycin: Healthy adults who will recieve one administration of 500 mg of Seromycin prior to the start of the study.
  Interventions: Drug: Seromycin
- Placebo: Healthy adults who will receive one administration of a placebo pill prior to the start of the study.

INTERVENTIONS:
Drug: Seromycin — 250 mg versus 500 mg versus placebo effects on conditioned fear generalization
  Other Names: D-cycloserine
  Groups: 250 mg Seromycin; 500 mg Seromycin
Drug: Seromycin
  Groups: 250 mg Seromycin; 500 mg Seromycin

SUMMARY:
PROJECT SUMMARY:

PTSD is a debilitating psychiatric condition precipitated by exposure to extreme, or life threatening, trauma with an estimated lifetime prevalence between 8% and 9% in U.S. adults. One core symptom of PTSD is intense psychological distress in the presence of stimuli that "resemble" one or more aspects of the trauma experience (DSM-IV). This phenomenon referred to as stimulus generalization has received surprisingly little empirical testing in the context of clinical anxiety in general, and PTSD more specifically. The current proposal represents the first effort to study the neurobiology and pharmacology of this PTSD-relevant learning phenomenon across those with and without PTSD. The objective of this particular proposal is to apply fMRI and pharmacologic methods to: 1) identify brain mechanisms associated with generalization of conditioned fear and 2) examine the pharmacologic modifiability of levels of generalization using a partial agonist at the NMDA receptor complex (D-cycloserine) shown to increase discrimination of CS+ (danger cue) and CS- (safety cue) in animal studies.

DETAILED DESCRIPTION:
To fullfill the objectives of this application, a generalization paradigm has been designed and psychophysiologically validated in which 6 rings presented on a computer screen gradually increase in size. For half of participants the smallest ring is the conditioned stimulus paired with electric shock (CS+) and the largest is the unpaired stimulus (CS-), and for the other half of participants this is reversed. Activity in fear-related brain structures measured via fMRI are predicted to gradually decrease as the presented stimulus gradually becomes less similar to the CS+, forming a generalization slope or gradient. One central hypothesis of the current application is that DCS (Seromycin) will dose dependently increase the steepness of generalization gradients (i.e., reduce fear generalization). This study will include 3 groups of healthy adults recieving either 1) 500 mg Seromycin, 2) 250 mg Seromycin, or placebo only prior to acquisition of fear conditioning. Twenty four hours later, participants will return to complete an fMRI during which brain responses to the danger cue and stimuli resembling the danger cue will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between the ages of 18-55.

Exclusion Criteria:

1. Current or past Axis I psychiatric diagnosis as determined by self report
2. Current substance dependence or meet criteria for the six month period preceding testing.
3. Participants will be excluded if they have current or past medical illnesses, which place the participant at risk or confound the results of the study including:

   A) Past history of hypersensitivity to Seromycin B) Current or past epileptic disorders C) Current depression D) Current anxiety disorders E) Current or past psychotic disorders F) Current or past renal disease G) Excessive or concurrent use of alcohol

   a) Subjects who are unable to abstain from alcohol for 12 hours prior to testing and 2 days following testing will be excluded
4. Current use of psychoactive medications or medications that alter central-nervous-system function
5. Females who are pregnant or currently breast-feeding
6. Any metallic implants or objects above the knee, tattoos about the knee, or oral braces.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults between the ages of 18-55.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2013-01; Primary Completion 2015-10-01 (Actual); Study Completion 2015-10-01 (Actual)

PRIMARY OUTCOMES:
fMRI (BOLD) responses | 1/1/13-6/1/14
  fMRI (BOLD) responses

SECONDARY OUTCOMES:
Behavioral assessments of perceived danger | up to three years
  Behavioral assessments of perceived danger

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Lissek, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of MInnesota, Minneapolis, Minnesota, United States